CLINICAL TRIAL: NCT03176823
Title: Remote Ischemic Conditioning as a Treatment for Traumatic Brain Injury: a Prospective Randomized Controlled Trial.
Brief Title: Remote Ischemic Conditioning as a Treatment for Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Defence Research and Development Canada (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RIC in TBI
Record Dates: First submitted 2017-05-15; First posted 2017-06-06 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Traumatic Brain Injury; Trauma, Nervous System; Reperfusion Injury; Ischemia, Brain
Keywords: Brain injury; Remote ischemic conditioning (RIC); Trauma; Biomarkers
MeSH Terms: conditions — Brain Injuries, Traumatic; Trauma, Nervous System; Reperfusion Injury; Brain Ischemia; Brain Injuries; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This trial is a prospective double-blind parallel cohort study of patients undergoing either standard of care plus placebo (sham-RIC) or standard treatment plus a single session of upper extremity remote ischemic conditioning.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: While it is not technically possible to mask participants to the application of RIC versus sham therapies, all participants in this trial by design will be intubated in an intensive care unit with severe traumatic brain injury; it is improbable that our inability to mask the patients will compromise outcomes or induce bias as patients are unlikely to have consciousness or memory of the therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Sham Comparator): Control-arm patients will be treated with standard "Best Practice" management of traumatic brain injury, with the addition of sham-RIC. The sham intervention will use a purpose-built device which will visually and audibly mimic a functional RIC device, with the key distinction being non-inflation of the arm cuff with resultant non-occlusion and no induced ischemia. To mask patient enrollment, all patients in both study arms will have the arm and RIC device draped in an opaque sheet so that the extremity distal to the RIC device are not visible to medical staff during the period of intervention.
  Interventions: Other: Best Practice Management of Traumatic Brain Injury
- RIC Arm (Experimental): The RIC treatment will be applied with a purpose-built commercial RIC device which will aid in standardizing dose and delivery. Therapeutic RIC will be provided by the CellAegis Technologies autoRIC device on an upper extremity. As with the control cohort, this cohort will undergo complete extremity draping.
  Interventions: Device: CellAegis Technologies autoRIC device; Other: Best Practice Management of Traumatic Brain Injury

INTERVENTIONS:
Device: CellAegis Technologies autoRIC device — The autoRIC device from CellAegis technologies will be applied as per the manufacturer's instructions on an upper extremity. The device will automatically inflate and deflate a blood pressure cuff to supra-systolic blood pressures, maintaining an occlusive pressure for a period of five minutes, followed by five minutes of re-perfusion with cuff deflation, completing a ten minute cycle. This cycle will repeat four times for a cumulative total of twenty minutes of occlusive conditioning over forty minutes of intervention time.
  Other Names: Remote Ischemic Conditioning
  Arms: RIC Arm
Other: Best Practice Management of Traumatic Brain Injury — Standard treatment of TBI in a dedicated trauma-neuro intensive care unit will include a tiered management strategy corresponding to many published treatment algorithms, including the American College of Surgeons Trauma Quality Improvement Program (ACS TQIP) guidelines for the management of intra-cranial hypertension. Standard practice without limitations will be applied to both cohorts of patients in this study.

SUMMARY:
The prevention of secondary brain injury is a primary goal in treating patients with severe traumatic brain injury (TBI). Secondary brain injury results from tissue ischemia induced by increased vascular resistance in the at-risk brain tissue due to compression by traumatic hematomas, and development of cytotoxic and vasogenic tissue edema. While traumatic hematomas may be managed surgically, cytotoxic and vasogenic edema with resulting perfusion impairment perpetuates brain ischemia and injury. Animal models suggest that remote ischemic conditioning (RIC) can reverse these effects and improve perfusion. Based on these findings it is hypothesized that RIC will exert beneficial effects on TBI in man, thereby representing a new therapeutic strategy for severe TBI.

Patients presenting to our institution suffering from severe TBI will be considered for enrollment. Eligible patients will have sustained a blunt, severe TBI (defined by Glasgow Coma Scale <8) with associated intra-cranial hematoma(s) not requiring immediate surgical decompression, with admission to an intensive care unit and insertion of an intra-cranial pressure monitor. Patients will be randomized to RIC versus sham-RIC intervention cohorts. RIC interventions will be performed using an automated device on the upper extremity delivering 20 cumulative minutes of limb ischemia in a single treatment session. The planned enrollment is a cohort of 40 patients.

Outcomes of this study will include multiple domains. Our primary outcome will include serial assessments of validated serum biomarkers of neuronal injury and systemic inflammation. Secondary outcomes will include descriptions of the clinical course of each patient, radiologic assessment of brain perfusion, and neurocognitive and psychological assessment post-discharge.

If clinical outcomes are improved using RIC, this study would support RIC as a novel treatment for TBI. Its advantages include safety and simplicity and, requiring no specialized equipment, its ability to be used in any environment including pre-hospital settings or in austere theatres. The investigators anticipate that TBI patients treated with RIC will have improved clinical, biochemical, and neuropsychological outcomes compared to standard treatment protocols.

DETAILED DESCRIPTION:
Traumatic brain injury is a leading cause of morbidity and mortality in victims of blunt trauma, leading to a tremendous economic cost, chronic neuropsychological sequelae and productive years of life lost. Treatment of inoperable primary brain injury consists largely of supportive care to support natural healing and prevention or reduction of secondary insults (1).

Many of the phenomena of secondary injury are related to ischemic sequelae of injury progression. Brain parenchymal edema increases both regional and global intra-cranial pressures, decreasing perfusion pressure, resulting in impaired perfusion, an oxygen debt, and ischemic injury (2). Local compression from traumatic hematomas may act in concert with edema to further impair perfusion. One strategy that has been successfully employed in the treatment of other ischemic insults is an intervention known as "remote ischemic conditioning" (RIC). RIC is felt to induce systemic responses which promote physiologic adaptations to moderate ischemia and minimize the impact of subsequent ischemic insults. Because these effects are systemic, extremity ischemic conditioning may impact brain injury. In the setting of TBI, where all patients carry a risk of ischemic secondary injury, early intervention with RIC may minimize the harm of secondary ischemic insults and improve outcomes.

The systemic effects of RIC have been demonstrated in a variety of organ systems and mechanisms of ischemia. Application of RIC has demonstrable benefits in preventing ischemia-induced organ dysfunction in insults to the heart (3-6), kidneys (7,8), and ocular organ systems (9). Our recent work has demonstrated its benefit in preventing organ injury following hemorrhagic shock (10). The technique has also demonstrated promise in reducing brain injury secondary to stroke or neurosurgical trauma (11-13).

Ischemic conditioning of brain injuries has proven benefits in animal models. Limb preconditioning reduces toxic oxygen free radicals, reduces neuronal apoptosis, reduces intra-cranial inflammation, improves integrity of the blood-brain barrier, and reduces brain parenchymal edema (14,15). RIC also improves microvascular perfusion to ischemic tissues which, in the brain, may reduce secondary injury by promoting perfusion to the at-risk injured brain (16). Even when performed after the intra-cranial trauma in a "post-conditioning" model, limb ischemic conditioning is associated with decreased apoptosis, decreased edema, and decreased brain infarction volumes (17,18). A single recent trial of RIC in human TBI patients showed a decrease in serum biomarkers of central nervous system (CNS) injury in the conditioned cohort (19).

Given the promising findings of the remote ischemic conditioning technique in reducing biomarkers of intra-cranial inflammation, an assessment of the clinical effectiveness of post-traumatic remote ischemic conditioning in modifying the outcomes of patients with isolated severe traumatic brain injuries is warranted.

Outcomes of this proposed prospective, randomized controlled trial will fall into the following validated categories:

1. Biomarkers of neuronal injury and systemic inflammation (20-28)
2. Radiologic evidence of improved acute- and delayed-phase perfusion (29-33)
3. Clinical course in hospital from admission to discharge
4. Neurocognitive and neuropsychological outcomes, 6 month follow-up (34-46)

The known physiologic effects of RIC are theoretically beneficial to patients suffering severe TBI who are at risk of clinical deterioration due to secondary injury. By mitigating the effects of inflammation and edema and improving microvascular perfusion, at-risk brain tissue may be salvaged and thus patient outcomes improved. This theory is supported by the existing evidence and a well-planned selection of outcome measures including biochemical, clinical, and radiographic outcomes may demonstrate the benefits of RIC in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Severe blunt traumatic brain injury presenting to St Michael's Hospital within 48 hours of trauma
* Glasgow Coma Scale (GCS) less than or equal to 12
* Presence on CT Scan of intra-cranial hematoma which adequately explains level of consciousness (epidural, subdural, subarachnoid hematomae)
* Able to undergo intervention within 48 hours of trauma

Exclusion Criteria:

* Age <18 years
* Lack of informed consent or withdrawal of consent, provided by legal substitute decision maker
* Unknown timing of trauma
* Unable to safely undergo ischemic conditioning of the upper extremity due to major trauma, previous surgery, known vascular disease or previous radiation treatment
* Acute significant injury (those injuries which in isolation would require admission to hospital) outside the head and neck region
* Pre-hospital therapeutic anticoagulation or anti-platelet agent use
* Surgical intervention within 12 hours of presentation to hospital, excluding pressure monitor insertion
* Patient death within 24 hours of admission
* Pre-intervention insertion of intra-cranial pressure monitor, as surgical trauma may influence biomarker measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Neuron Specific Enolase (NSE) - biomarker | Admission (0 hours), 6 hours, 24 hours, 48 hours, and 72 hours
  Plasma concentration measured by measured by enzyme-linked immunosorbent ELISA and multiplex platform at all time points specified below.
S100A12 - biomarker | Admission (0 hours), 6 hours, 24 hours, 48 hours, and 72 hours
  Plasma concentration measured by measured by enzyme-linked immunosorbent ELISA and multiplex platform at all time points specified below.
Calcium Binding Protein Beta (S100B) - biomarker | Admission (0 hours), 6 hours, 24 hours, 48 hours, and 72 hours
  Plasma concentration measured by measured by enzyme-linked immunosorbent ELISA and multiplex platform at all time points specified below.
Glial Fibrillary Acidic Protein (GFAP) - biomarker | Admission (0 hours), 6 hours, 24 hours, 48 hours, and 72 hours
  Plasma concentration measured by measured by enzyme-linked immunosorbent ELISA and multiplex platform at all time points specified below.
Monocyte Chemoattractant Protein (MCP1) - biomarker | Admission (0 hours), 6 hours, 24 hours, 48 hours, and 72 hours
  Plasma concentration measured by measured by enzyme-linked immunosorbent ELISA and multiplex platform at all time points specified below.
Epinephrine - biomarker | Admission (0 hours), 6 hours, 24 hours, 48 hours, and 72 hours
  Plasma concentration measured by measured by enzyme-linked immunosorbent ELISA and multiplex platform at all time points specified below.
Norepinephrine - biomarker | Admission (0 hours), 6 hours, 24 hours, 48 hours, and 72 hours
  Plasma concentration measured by measured by enzyme-linked immunosorbent ELISA and multiplex platform at all time points specified below.
Interleukin 10 (IL10) - biomarker | Admission (0 hours), 6 hours, 24 hours, 48 hours, and 72 hours
  Plasma concentration measured by measured by enzyme-linked immunosorbent ELISA and multiplex platform at all time points specified below.
Interleukin 1 Beta (IL1B) - biomarker | Admission (0 hours), 6 hours, 24 hours, 48 hours, and 72 hours
  Plasma concentration measured by measured by enzyme-linked immunosorbent ELISA and multiplex platform at all time points specified below.
Tumor Necrosis Factor Alpha (TNF Alpha) - biomarker | Admission (0 hours), 6 hours, 24 hours, 48 hours, and 72 hours
  Plasma concentration measured by measured by enzyme-linked immunosorbent ELISA and multiplex platform at all time points specified below.
International Normalized Ratio (INR) - standard lab test. | Admission (0 hours), 6 hours, 24 hours, 48 hours, and 72 hours
  Standard coagulation parameter, to be measured at all time points specified below.
Prothrombin Time (PTT) - standard lab test. | Admission (0 hours), 6 hours, 24 hours, 48 hours, and 72 hours
  Standard coagulation parameter, to be measured at all time points specified below
Rotational Thromboelastometry (ROTEM), standard lab test. | Admission (0 hours), 6 hours, 24 hours, 48 hours, and 72 hours
  ROTEM coagulation assessment using the commercial ROTEM device traditionally used for the assessment of trauma-induced coagulopathy, to be measured at all time points specified below

SECONDARY OUTCOMES:
Cerebral vascular perfusion, acute | 24 hours
  Patients will undergo Arterial Spin Loading Functional Magnetic Resonance Imaging (fMRI) at 72 hours post-RIC to quantify blood flow to the acutely ischemic brain parenchyma.
Intracranial Pressure (ICP) measurement, first 24 hours | 24 hours
  The number of episodes of ICP >20 mmHg, measured in 15 minute increments, over the first 24 hours.
Intracranial Pressure (ICP) measurement, 24-96 hours | 24 hours, 96 hours
  The number of episodes of ICP >20 mmHg, measured in 15 minute increments, over 24-96 hours.
Escalation along an established care algorithm | 12 months
  Patient care interventions will be plotted against the Tier 1, Tier 2, and Tier 3 categories of interventions described by the American College of Surgeons Trauma Quality Improvement Program (ACS TQIP) guidelines for the management of traumatic intracranial hypertension.
Mortality beyond 12 hours post-admission | 12 months
  Patient deaths occurring in the first 12 hours will result in patient-exclusion as it is unlikely that these patients would have had different outcomes regardless of treatment strategies.
Incidence of surgical decompression beyond 12 hours post-admission | 12 months
  Patient progression to need for definitive surgery occurring in the first 12 hours will result in patient-exclusion as it is unlikely that these patients would have had different outcomes regardless of treatment strategies.
Hospital length of stay, number of days | 12 months
  Number of continuous calendar days or partial calendar days admitted to an acute-care hospital.
Intensive Care Unit length of stay, number of days | 2 months
  Number of continuous calendar days or partial calendar days admitted to an intensive-care unit.
Total duration of mechanical ventilation, number of days | 2 months
  Number of calendar days or partial calendar days including treatment with invasive ventilation.
Destination of discharge | 12 months
  Home (functionally independent), rehabilitation facility, or chronic care facility
Glasgow Outcomes Scale, Extended (GOSE) - neurocognitive test | discharge, 3 months, 6 months, and 12 months
  The GOSE scale assessing neurocognitive function will be assessed on hospital, discharge, at three months post-discharge, and at 6 and 12 months post-discharge.
Disability Rating Scale (DRS) - neurocognitive function rating | discharge, 3 months, 6 months, and 12 months
  The DRS scale assessing neurocognitive function will be assessed on hospital discharge, at three months post-discharge, and at 6 and 12 months post-discharge.
Patient Health Questionnaire 9th edition (PHQ-9) - neurological - self assessment | discharge, 3, 6, and 12 months
  The PHQ-9 screen for mental health disorders will be assessed on hospital discharge, at three months post-discharge, and at 6 and 12 months post-discharge.
Posttraumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual of Mental Disorders 5th edition (PCL-5) - neurological - self assessment | discharge, 3 months, 6 months, and 12 months
  The PCL-5 screen for Post-Traumatic Stress Disorder will be assessed on hospital discharge, at three months post-discharge, and at 6 and 12 months post-discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Ori D Rotstein, MD, Principal Investigator — Unity Health Toronto - St. Michael's hospital
Locations (1):
- St Michaels Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ACS TQIP Best Practices in the Management of Traumatic Brain Injury. 2015.
- [Background] Bouma GJ, Muizelaar JP, Choi SC, Newlon PG, Young HF. Cerebral circulation and metabolism after severe traumatic brain injury: the elusive role of ischemia. J Neurosurg. 1991 Nov;75(5):685-93. doi: 10.3171/jns.1991.75.5.0685. PMID 1919689
- [Background] Botker HE, Kharbanda R, Schmidt MR, Bottcher M, Kaltoft AK, Terkelsen CJ, Munk K, Andersen NH, Hansen TM, Trautner S, Lassen JF, Christiansen EH, Krusell LR, Kristensen SD, Thuesen L, Nielsen SS, Rehling M, Sorensen HT, Redington AN, Nielsen TT. Remote ischaemic conditioning before hospital admission, as a complement to angioplasty, and effect on myocardial salvage in patients with acute myocardial infarction: a randomised trial. Lancet. 2010 Feb 27;375(9716):727-34. doi: 10.1016/S0140-6736(09)62001-8. PMID 20189026
- [Background] Sloth AD, Schmidt MR, Munk K, Kharbanda RK, Redington AN, Schmidt M, Pedersen L, Sorensen HT, Botker HE; CONDI Investigators. Improved long-term clinical outcomes in patients with ST-elevation myocardial infarction undergoing remote ischaemic conditioning as an adjunct to primary percutaneous coronary intervention. Eur Heart J. 2014 Jan;35(3):168-75. doi: 10.1093/eurheartj/eht369. Epub 2013 Sep 12. PMID 24031025
- [Background] Pei H, Wu Y, Wei Y, Yang Y, Teng S, Zhang H. Remote ischemic preconditioning reduces perioperative cardiac and renal events in patients undergoing elective coronary intervention: a meta-analysis of 11 randomized trials. PLoS One. 2014 Dec 31;9(12):e115500. doi: 10.1371/journal.pone.0115500. eCollection 2014. PMID 25551671
- [Background] Davies WR, Brown AJ, Watson W, McCormick LM, West NE, Dutka DP, Hoole SP. Remote ischemic preconditioning improves outcome at 6 years after elective percutaneous coronary intervention: the CRISP stent trial long-term follow-up. Circ Cardiovasc Interv. 2013 Jun;6(3):246-51. doi: 10.1161/CIRCINTERVENTIONS.112.000184. Epub 2013 May 21. PMID 23696599
- [Background] Er F, Nia AM, Dopp H, Hellmich M, Dahlem KM, Caglayan E, Kubacki T, Benzing T, Erdmann E, Burst V, Gassanov N. Ischemic preconditioning for prevention of contrast medium-induced nephropathy: randomized pilot RenPro Trial (Renal Protection Trial). Circulation. 2012 Jul 17;126(3):296-303. doi: 10.1161/CIRCULATIONAHA.112.096370. Epub 2012 Jun 26. PMID 22735306
- [Background] Zarbock A, Schmidt C, Van Aken H, Wempe C, Martens S, Zahn PK, Wolf B, Goebel U, Schwer CI, Rosenberger P, Haeberle H, Gorlich D, Kellum JA, Meersch M; RenalRIPC Investigators. Effect of remote ischemic preconditioning on kidney injury among high-risk patients undergoing cardiac surgery: a randomized clinical trial. JAMA. 2015 Jun 2;313(21):2133-41. doi: 10.1001/jama.2015.4189. PMID 26024502
- [Background] Liu X, Sha O, Cho EY. Remote ischemic postconditioning promotes the survival of retinal ganglion cells after optic nerve injury. J Mol Neurosci. 2013 Nov;51(3):639-46. doi: 10.1007/s12031-013-0036-2. Epub 2013 Jun 5. PMID 23733254
- [Background] Leung CH, Caldarone CA, Wang F, Venkateswaran S, Ailenberg M, Vadasz B, Wen XY, Rotstein OD. Remote Ischemic Conditioning Prevents Lung and Liver Injury After Hemorrhagic Shock/Resuscitation: Potential Role of a Humoral Plasma Factor. Ann Surg. 2015 Jun;261(6):1215-25. doi: 10.1097/SLA.0000000000000877. PMID 25185480
- [Background] DAHL NA, BALFOUR WM. PROLONGED ANOXIC SURVIVAL DUE TO ANOXIA PRE-EXPOSURE: BRAIN ATP, LACTATE, AND PYRUVATE. Am J Physiol. 1964 Aug;207:452-6. doi: 10.1152/ajplegacy.1964.207.2.452. No abstract available. PMID 14205366
- [Background] Kitagawa K, Matsumoto M, Tagaya M, Hata R, Ueda H, Niinobe M, Handa N, Fukunaga R, Kimura K, Mikoshiba K, et al. 'Ischemic tolerance' phenomenon found in the brain. Brain Res. 1990 Sep 24;528(1):21-4. doi: 10.1016/0006-8993(90)90189-i. PMID 2245337
- [Background] Chen J, Graham SH, Zhu RL, Simon RP. Stress proteins and tolerance to focal cerebral ischemia. J Cereb Blood Flow Metab. 1996 Jul;16(4):566-77. doi: 10.1097/00004647-199607000-00006. PMID 8964795
- [Background] Wei D, Ren C, Chen X, Zhao H. The chronic protective effects of limb remote preconditioning and the underlying mechanisms involved in inflammatory factors in rat stroke. PLoS One. 2012;7(2):e30892. doi: 10.1371/journal.pone.0030892. Epub 2012 Feb 8. PMID 22347410
- [Background] Wang Y, Ge P, Yang L, Wu C, Zha H, Luo T, Zhu Y. Protection of ischemic post conditioning against transient focal ischemia-induced brain damage is associated with inhibition of neuroinflammation via modulation of TLR2 and TLR4 pathways. J Neuroinflammation. 2014 Jan 24;11:15. doi: 10.1186/1742-2094-11-15. PMID 24460643
- [Background] Schoen M, Rotter R, Gierer P, Gradl G, Strauss U, Jonas L, Mittlmeier T, Vollmar B. Ischemic preconditioning prevents skeletal muscle tissue injury, but not nerve lesion upon tourniquet-induced ischemia. J Trauma. 2007 Oct;63(4):788-97. doi: 10.1097/01.ta.0000240440.85673.fc. PMID 18090007
- [Background] Ren C, Gao M, Dornbos D 3rd, Ding Y, Zeng X, Luo Y, Ji X. Remote ischemic post-conditioning reduced brain damage in experimental ischemia/reperfusion injury. Neurol Res. 2011 Jun;33(5):514-9. doi: 10.1179/016164111X13007856084241. PMID 21669121
- [Background] Liu X, Zhao S, Liu F, Kang J, Xiao A, Li F, Zhang C, Yan F, Zhao H, Luo M, Luo Y, Ji X. Remote ischemic postconditioning alleviates cerebral ischemic injury by attenuating endoplasmic reticulum stress-mediated apoptosis. Transl Stroke Res. 2014 Dec;5(6):692-700. doi: 10.1007/s12975-014-0359-5. Epub 2014 Jul 22. PMID 25043802
- [Background] Joseph B, Pandit V, Zangbar B, Kulvatunyou N, Khalil M, Tang A, O'Keeffe T, Gries L, Vercruysse G, Friese RS, Rhee P. Secondary brain injury in trauma patients: the effects of remote ischemic conditioning. J Trauma Acute Care Surg. 2015 Apr;78(4):698-703; discussion 703-5. doi: 10.1097/TA.0000000000000584. PMID 25742251
- [Background] Di Battista AP, Buonora JE, Rhind SG, Hutchison MG, Baker AJ, Rizoli SB, Diaz-Arrastia R, Mueller GP. Blood Biomarkers in Moderate-To-Severe Traumatic Brain Injury: Potential Utility of a Multi-Marker Approach in Characterizing Outcome. Front Neurol. 2015 May 26;6:110. doi: 10.3389/fneur.2015.00110. eCollection 2015. PMID 26074866
- [Background] Lewis LM, Schloemann DT, Papa L, Fucetola RP, Bazarian J, Lindburg M, Welch RD. Utility of Serum Biomarkers in the Diagnosis and Stratification of Mild Traumatic Brain Injury. Acad Emerg Med. 2017 Jun;24(6):710-720. doi: 10.1111/acem.13174. Epub 2017 May 18. PMID 28170122
- [Background] Thelin EP, Nelson DW, Bellander BM. A review of the clinical utility of serum S100B protein levels in the assessment of traumatic brain injury. Acta Neurochir (Wien). 2017 Feb;159(2):209-225. doi: 10.1007/s00701-016-3046-3. Epub 2016 Dec 12. PMID 27957604
- [Background] Semple BD, Bye N, Rancan M, Ziebell JM, Morganti-Kossmann MC. Role of CCL2 (MCP-1) in traumatic brain injury (TBI): evidence from severe TBI patients and CCL2-/- mice. J Cereb Blood Flow Metab. 2010 Apr;30(4):769-82. doi: 10.1038/jcbfm.2009.262. Epub 2009 Dec 23. PMID 20029451
- [Background] Vos PE, Jacobs B, Andriessen TM, Lamers KJ, Borm GF, Beems T, Edwards M, Rosmalen CF, Vissers JL. GFAP and S100B are biomarkers of traumatic brain injury: an observational cohort study. Neurology. 2010 Nov 16;75(20):1786-93. doi: 10.1212/WNL.0b013e3181fd62d2. PMID 21079180
- [Background] Vos PE, Lamers KJ, Hendriks JC, van Haaren M, Beems T, Zimmerman C, van Geel W, de Reus H, Biert J, Verbeek MM. Glial and neuronal proteins in serum predict outcome after severe traumatic brain injury. Neurology. 2004 Apr 27;62(8):1303-10. doi: 10.1212/01.wnl.0000120550.00643.dc. PMID 15111666
- [Background] Brohi K, Singh J, Heron M, Coats T. Acute traumatic coagulopathy. J Trauma. 2003 Jun;54(6):1127-30. doi: 10.1097/01.TA.0000069184.82147.06. PMID 12813333
- [Background] Stein SC, Smith DH. Coagulopathy in traumatic brain injury. Neurocrit Care. 2004;1(4):479-88. doi: 10.1385/NCC:1:4:479. PMID 16174954
- [Background] Schochl H, Solomon C, Traintinger S, Nienaber U, Tacacs-Tolnai A, Windhofer C, Bahrami S, Voelckel W. Thromboelastometric (ROTEM) findings in patients suffering from isolated severe traumatic brain injury. J Neurotrauma. 2011 Oct;28(10):2033-41. doi: 10.1089/neu.2010.1744. Epub 2011 Sep 23. PMID 21942848
- [Background] Shen Y, Kou Z, Kreipke CW, Petrov T, Hu J, Haacke EM. In vivo measurement of tissue damage, oxygen saturation changes and blood flow changes after experimental traumatic brain injury in rats using susceptibility weighted imaging. Magn Reson Imaging. 2007 Feb;25(2):219-27. doi: 10.1016/j.mri.2006.09.018. Epub 2006 Nov 28. PMID 17275617
- [Background] Kim J, Whyte J, Patel S, Avants B, Europa E, Wang J, Slattery J, Gee JC, Coslett HB, Detre JA. Resting cerebral blood flow alterations in chronic traumatic brain injury: an arterial spin labeling perfusion FMRI study. J Neurotrauma. 2010 Aug;27(8):1399-411. doi: 10.1089/neu.2009.1215. PMID 20528163
- [Background] Hunter JV, Wilde EA, Tong KA, Holshouser BA. Emerging imaging tools for use with traumatic brain injury research. J Neurotrauma. 2012 Mar 1;29(4):654-71. doi: 10.1089/neu.2011.1906. Epub 2011 Oct 17. PMID 21787167
- [Background] Lopez-Aguilera F, Plateo-Pignatari MG, Biaggio V, Ayala C, Seltzer AM. Hypoxic preconditioning induces an AT2-R/VEGFR-2(Flk-1) interaction in the neonatal brain microvasculature for neuroprotection. Neuroscience. 2012 Aug 2;216:1-9. doi: 10.1016/j.neuroscience.2012.04.070. Epub 2012 May 6. PMID 22569153
- [Background] Thompson WH, Thelin EP, Lilja A, Bellander BM, Fransson P. Functional resting-state fMRI connectivity correlates with serum levels of the S100B protein in the acute phase of traumatic brain injury. Neuroimage Clin. 2016 May 9;12:1004-1012. doi: 10.1016/j.nicl.2016.05.005. eCollection 2016. PMID 27995066
- [Background] Struchen MA, Hannay HJ, Contant CF, Robertson CS. The relation between acute physiological variables and outcome on the Glasgow Outcome Scale and Disability Rating Scale following severe traumatic brain injury. J Neurotrauma. 2001 Feb;18(2):115-25. doi: 10.1089/08977150150502569. PMID 11229706
- [Background] Hall K, Cope DN, Rappaport M. Glasgow Outcome Scale and Disability Rating Scale: comparative usefulness in following recovery in traumatic head injury. Arch Phys Med Rehabil. 1985 Jan;66(1):35-7. PMID 3966866
- [Background] Levin HS, Boake C, Song J, Mccauley S, Contant C, Diaz-Marchan P, Brundage S, Goodman H, Kotrla KJ. Validity and sensitivity to change of the extended Glasgow Outcome Scale in mild to moderate traumatic brain injury. J Neurotrauma. 2001 Jun;18(6):575-84. doi: 10.1089/089771501750291819. PMID 11437080
- [Background] Gouvier WD, Blanton PD, LaPorte KK, Nepomuceno C. Reliability and validity of the Disability Rating Scale and the Levels of Cognitive Functioning Scale in monitoring recovery from severe head injury. Arch Phys Med Rehabil. 1987 Feb;68(2):94-7. PMID 3813863
- [Background] McMillan T, Wilson L, Ponsford J, Levin H, Teasdale G, Bond M. The Glasgow Outcome Scale - 40 years of application and refinement. Nat Rev Neurol. 2016 Aug;12(8):477-85. doi: 10.1038/nrneurol.2016.89. Epub 2016 Jul 15. PMID 27418377
- [Background] Seel RT, Kreutzer JS, Rosenthal M, Hammond FM, Corrigan JD, Black K. Depression after traumatic brain injury: a National Institute on Disability and Rehabilitation Research Model Systems multicenter investigation. Arch Phys Med Rehabil. 2003 Feb;84(2):177-84. doi: 10.1053/apmr.2003.50106. PMID 12601647
- [Background] Kreutzer JS, Seel RT, Gourley E. The prevalence and symptom rates of depression after traumatic brain injury: a comprehensive examination. Brain Inj. 2001 Jul;15(7):563-76. doi: 10.1080/02699050010009108. PMID 11429086
- [Background] Warren AM, Boals A, Elliott TR, Reynolds M, Weddle RJ, Holtz P, Trost Z, Foreman ML. Mild traumatic brain injury increases risk for the development of posttraumatic stress disorder. J Trauma Acute Care Surg. 2015 Dec;79(6):1062-6. doi: 10.1097/TA.0000000000000875. PMID 26488326
- [Background] Schneiderman AI, Braver ER, Kang HK. Understanding sequelae of injury mechanisms and mild traumatic brain injury incurred during the conflicts in Iraq and Afghanistan: persistent postconcussive symptoms and posttraumatic stress disorder. Am J Epidemiol. 2008 Jun 15;167(12):1446-52. doi: 10.1093/aje/kwn068. Epub 2008 Apr 17. PMID 18424429
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250